CLINICAL TRIAL: NCT04375553
Title: Effects of a Program of Aerobic Exercise on the Profile of Intestinal Microbiota and Cardiovascular Markers in Patients With Chronic Kidney Disease
Brief Title: Aerobic Exercise in Patients With CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Denise Mafra 5
Record Dates: First submitted 2019-04-25; First posted 2020-05-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Active Comparator): Intradialytic aerobic exercise, 3 times a week, for 12 weeks.
  Interventions: Other: Aerobic exercise
- Non-exercise group (No Intervention): Without intradialytic aerobic exercise for 12 weeks.

INTERVENTIONS:
Other: Aerobic exercise — Intradialytic aerobic exercise
  Arms: Exercise group

SUMMARY:
Patients with chronic kidney disease (CKD), especially those who are on dialysis, have a high prevalence of cardiovascular mortality and among the risk factors; inflammation and oxidative stress stand out. Furthermore, recently this scenario, beyond those alterations found in these patients, it has been suggested that the imbalance gut microbiota might be a new factor of cardiovascular risk. Some treatment strategies have been studied in order to modulate the gut microbiota and inflammation, such as the implementation of exercise programs. However, the effects of exercise on the modulation of the gut microflora and inflammation have not been evaluated in these patients. The aim of this project is to investigate possible changes in gut microbiota, levels of uremic toxins and inflammatory and cardiovascular markers in CKD patients on hemodialysis, after application of a training program with aerobic exercise.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) patients on hemodialysis (HD) patients present reduced functional capacity to approximately 50% and uremic myopathy and disuse atrophy have a significant impact on the functional capacity of these patients (Johansen, 1999; Parsons, 2006).

There are several physical exercise benefits for CKD patients, such as improved ability to perform exercises, increase of strength, quality of life and improve the maximal oxygen consumption (VO2MÁX), which contributes to the improvement of cardiovascular aspects (Johansen, 2007; Johansen, 2005; Heiwe, 2014). In fact, CKD patients who practice regular exercise have a higher survival rate (O'Hare et al., 2003).

In addition, some mechanisms regarding anti-inflammatory effects of the exercises has been proposed, such as: reduction of visceral fat which decreases the secretion of pro-inflammatory cytokines, increased production and release of anti-inflammatory cytokines from muscle contraction and reduced expression of Toll-like receptors (TLRs) in monocytes and macrophages, which decreases the pro-inflammatory response (Petersen & Pedersen, 2005; Gleeson et al., 2006).

In parallel, during exercises like running or cycling, there is an increase in capillary surface area, with opening of capillaries previously inactive, consequently increasing exchange of substances between the blood and the tissues. Thus, physical exercise could result in a greater flux of urea and associated toxins from tissue to vascular compartment, improving the efficiency of dialysis (Parsons et al., 2006; Guyton E Hall, 2017). According KDOQI (Kidney Disease Outcomes Quality Initiative), Kt/V, a measure of urea clearance, is the most frequently applied measure of the delivered dialysis dose and reflects the dialyzer effect on patient survival (KDOQI, 2015).

Despite results showing the benefits of exercise to CKD patients, they are poorly prescribed, remaining a challenge in clinical practice and high rates of physical inactivity are observed in these patients (Williams et al., 2014; Barcellos, 2018).

Some gaps still need to be filled regarding the not yet known effect of physical exercise on a number of clinical factors, thus allowing more specific and objective recommendations (Williams et al., 2014). In this context, the present study aims to verify the effects of 12-week supervised and individualized intradialytic bicycle ergometer exercise on the adequacy of dialysis, inflammatory markers and functional capacity of HD patients.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary men and women between the ages of 18 and 60;
* patients with hemodialysis only with vascular access arteriovenous fistula who have been in dialysis for more than 6 months
* patients with hemoglobin levels greater than 10 mg / dL.

Exclusion Criteria:

* Patients taking catabolizing drugs, vitamin supplements, antioxidants, probiotics, prebiotics, symbiotics and antibiotics;
* patients with autoimmune, infectious, cancer, AIDS,
* patients with clinically unstable diseases (AMI less than 1 year, unstable angina, atrial fibrillation, significant cardiac arrhythmia and acute disease in the last month)
* patients with frequent hypotension during dialysis
* patients with chronic obstructive pulmonary disease and glycemic lability;
* incapacitated to perform exercise (amputation without prosthesis);
* musculoskeletal pain at rest or with minimal physical activity,
* inability to sit or walk without assistance,
* dyspnoea at rest or at slight exertion (NYHA III and IV).
* impediment to completing the proposed exercise protocol (travel, imminent renal transplantation).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Inflammatory biomarkers | 12 weeks
  Get blood samples to evaluate changes in the expression of transcription factors (nuclear factor erythroid 2-related factor 2 and Nuclear Factor-kB) that modulate inflammation.
Uremic toxins | 12 weeks
  Evaluation of P-Cresyl Sulfate, Indoxyl Sulfate (IS), Indole 3-Acetic Acid, Trimethyl N-oxide (TMAO) and lipopolysaccharides (LPSs).

CONTACTS AND LOCATIONS:
Overall Officials: Denise Mafra, PhD, Principal Investigator — Federal university fluminense
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brito JS, Borges NA, Reis DCMV, Silva GSD, Fonseca LDS, Ribeiro MMF, Chermut TR, Moura MC, Oliveira LC, Paiva BR, Cardozo LF, Capistrano ESM, Mafra D. Effects of intradialytic bicycle ergometer exercise on transcription factors NF-kB and Nrf2 in patients with chronic kidney disease: A randomized crossover clinical trial. J Bodyw Mov Ther. 2024 Oct;40:1492-1501. doi: 10.1016/j.jbmt.2024.08.003. Epub 2024 Aug 8. PMID 39593477
- [Derived] Brito JS, Reis D, Silva G, Fonseca L, Ribeiro M, Chermut T, Oliveira L, Borges NA, Ribeiro-Alves M, Mafra D. Bicycle ergometer exercise during hemodialysis and its impact on quality of life, aerobic fitness and dialysis adequacy: A pilot study. Complement Ther Clin Pract. 2022 Nov;49:101669. doi: 10.1016/j.ctcp.2022.101669. Epub 2022 Sep 17. PMID 36152526